CLINICAL TRIAL: NCT06566560
Title: Cost-savings and Environmental Impact Obtained From Redispensing Unused Oral Anticancer Drugs
Brief Title: The ROAD 2.0 to Sustainable Medication Use: Redispensing Unused Oral Anticancer Drugs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-7049; 111109 (Other: PaNaMa)
Record Dates: First submitted 2024-08-06; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Cancer; Oncology; Pharmacy; Drug Prescriptions
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other)
  Interventions: Other: redispensing oral anticancer drugs

INTERVENTIONS:
Other: redispensing oral anticancer drugs — Participants will receive oral anticancer drugs according to their regular prescriptions, distributed in the original manufacturer's package. Following the guideline, some oral anticancer drug (i.e. requiring temperature storage up to 25C degrees) will be supplemented with a validated temperature indicator (Timestrip Neo, customer configuration), enclosed with a seal bag. Patients are requested to return unused oral anticancer drugs to the outpatient pharmacy that distributed them.
  Pharmacy staff will assess the quality of returned oral anticancer drugs, applying the following criteria:
  1. the seal bag is unopened
  2. the drug package is unopend and undamaged
  3. the expiry date is ≥ 3 months
  4. the medication has not been stored outside the product label storage claim
  Oral anticancer drugs that meet all criteria are restocked, and consecutively redispensed to participants visiting the same outpatient pharmacy.

SUMMARY:
The goal of this prospective intervention study is to investigate the effectiveness of redispensing unused oral anticancer drugs.

The main questions it aims to answer are:

* What are the cost-savings of redispensing unused oral anticancer drugs?
* What is the environmental impact of redispensing unused oral anticancer drugs?

Researchers will compare redispensing unused oral anticancer drugs to the standard practice of disposal.

Participants will receive their oral anticancer drugs in a sealed bag with a temperature indicator if needed. They will be asked to return any unused oral anticancer drugs to the pharmacy during their next visit to the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages
* A clinical diagnosis of cancer using an oral anticancer drug that requires storage at room temperature according to the Summary of Product Characteristics (SmPC).

Exclusion Criteria:

* Patients that do not understand the Dutch or English language, in written or spoken.
* Patients receiving prescriptions that contain an amount of tablets that deviates from the regular package size, resulting in the pharmacy dispensing an opened package

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The environmental impact of redispensing unused oral anticancer drugs of verified quality compared to standard practice of disposal. | From date of first dispensing unit the date of last unused medication package returning to the pharmacy, assessed up to 16 months
  Environmental impact will be measured in CO2-eq
Cost-savings obtained by redispensing unused oral anticancer drugs of verified quality compared to standard practice of disposal. | From date of first dispensing unit the date of last unused medication package returning to the pharmacy, assessed up to 16 months.
  Cost savings will be measured in euros

SECONDARY OUTCOMES:
The proportion of usability of returned medication for redispensing and the reasons for quality disapproval. | From date of first dispensing unit the date of last unused medication package returning to the pharmacy, assessed up to 16 months
The proportion of returned unused oral anticancer drugs and reasons thereof. | From date of first dispensing unit the date of last unused medication package returning to the pharmacy, assessed up to 16 months
Patients' reasons for not wanting to participate in a redispensing program for oral anticancer drugs. | From date of first invitation to participate in the study until the end of the recruitment period, up to 8 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes